CLINICAL TRIAL: NCT01910077
Title: An Open Label, Randomized, Single Dose, Crossover Pivotal Bioequivalence Study of Tacrobell Capsule 1mg Versus Prograf Capsule 1mg in Healthy Subjects
Brief Title: Bioequivalence Study of Tacrobell Capsule 1mg to Prograf Capsule 1mg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Tacrobell_BE-1301
Record Dates: First submitted 2013-07-24; First posted 2013-07-29 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Immunosuppression
Keywords: tacrolimus; tacrobell capsule; prograf capsule; bioequivalence
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tacrobell capsule 1mg (Experimental): Tacrolimus 1mg / 1 capsule
  Interventions: Drug: Tacrobell capsule 1mg
- Prograf capsule 1mg (Active Comparator): Tacrolimus 1mg / 1 capsule
  Interventions: Drug: Prograf capsule 1mg

INTERVENTIONS:
Drug: Tacrobell capsule 1mg — 1 capsule, oral, over the period I&II(crossover)
  Arms: Tacrobell capsule 1mg
Drug: Prograf capsule 1mg — 1 capsule, oral, over the period I&II(crossover)
  Arms: Prograf capsule 1mg

SUMMARY:
The purpose of this study is to demonstrate bioequivalence between tacrobell capsule 1mg and prograf capsule 1mg.

DETAILED DESCRIPTION:
This will be an open label, randomized, single dose, 2-treatment, 2-period crossover study in healthy volunteers.Study treatments will be administered under fasting conditions.

Blood samples for the analysis of tacrolimus in blood will be obtained as follows: Predose(immediately prior to dosing), and at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours postdose.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent from prior to screening test
* Between 19 years and 55 years in healthy male subject
* Have not any congenital or chronic disease and medical symptoms
* Body mass index(BMI) of 18 to 30 and a total body weight ≥ 55kg
* Appropriate subject for the study judging from investigator

Exclusion Criteria:

* Evidence or history of clinically significant hepatic, renal, neurologic, immune system, respiratory system, endocrine
* Any condition possibly affecting drug absorption (e.g. gastrectomy)
* Subject with hypersensitivity to tacrolimus or any excipient
* Administration of cyclosporin or bosentan
* Administration of potassium-sparing diuretics
* Subject with hereditary diseases of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* SBP<90 mmHg or DBP<50 mmHg, SBP>150 mmHg or DBP>100 mmHg at least 3 minutes of rest
* A positive HBsAg, HCV Ab, HIV Ab, RPR
* AST, ALT > 1.5*upper limit of normal range at the screening test
* Subject with a history of drug abuse or a positive reaction for drug abuse at the screening test
* Taking ETC medicine including oriental medicine within 14days before the first hospitalization or taking OTC medicine, vitamin within 7days
* Use of any drugs known to significantly induce or inhibit drug-metabolizing enzymes within 30 days prior to initiation test
* Participating in a bioequivalence study or other clinical study within 3 month preceding the first hospitalization
* Blood donation or more within 2 month or component blood donation within 1 month prior to the first hospitalization
* Continued to be drinking(alcohol> 21 units/week, 1 unit=10g of pure alcohol) or during clinical trials can not be drunk
* Severe heavy smoker(cigarette> 10 cigarettes/day) during 3 months or can not be smoking during the clinical study
* Continued to be taking caffeine or can not be taken caffeine
* Continued to be taking grapefruit or can not be taken grapefruit
* Not use of contraception during the clinical study
* An impossible one who participates in the clinical trial by investigator's decision including for reason of laboratory test result

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-08; Primary Completion 2013-08 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
AUClast | At pre-dose (immediately prior to dosing) and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours postdese
  AUClast: Area under the blood concentration-time profile from time zero to the time of the last quantifiable concentration
Cmax | At pre-dose (immediately prior to dosing) and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours postdese
  Cmax: Maximum blood concentration

SECONDARY OUTCOMES:
AUCinf | At pre-dose (immediately prior to dosing) and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours postdose
  ACUinf: Area under the blood concentration-time profile from time zero extrapolated to infinite time
Tmax | At pre-dose (immediately prior to dosing) and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours postdose
  Tmax: Time for Cmax
T1/2 | At pre-dose (immediately prior to dosing) and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours postdose
  T1/2: Terminal elimination half-life
CL/F | At pre-dose (immediately prior to dosing) and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 6, 8, 12, 24, 48, 72 and 96 hours postdose
  CL/F: Apparent Clearance

CONTACTS AND LOCATIONS:
Overall Officials: Hyeong Ki Lee, MD, Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul national university hospital, Seoul, South Korea